CLINICAL TRIAL: NCT05017246
Title: A Randomized Trial Comparing Intrathecal Morphine and Intraoperative Lidocaine Infusion to Epidural Anesthesia With Postoperative PCA for Patients Undergoing Exploratory Laparotomy on the Gynecologic Oncology Service.
Brief Title: Comparing Intrathecal Morphine and Intraoperative Lidocaine Infusion to Epidural Anesthesia With Postoperative PCA for Patients Undergoing Exploratory Laparotomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202105007
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cancer Debulking; Enlarged Uterus; Fibroid Uterus; Adnexal Mass
Keywords: ERAS; Multi-modal anesthesia; Opioid consumption; Intrathecal; Epidural; Ileus
MeSH Terms: conditions — Leiomyoma; Ileus | interventions — Bupivacaine; Morphine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epidural bupivacaine with hydromorphone patient-controlled anesthesia (EPCA) (Active Comparator): * Standard of care at Washington University School of Medicine/Barnes-Jewish Hospital
  * Day of surgery: preoperative tylenol, gabapentin, celebrex, and epidural dosing per standard protocol.
  * Intraoperative: dexamethasone and epidural bupivacaine
  * Day of surgery postoperative: hydromorphone PCA, toradol, ibuprofen, tylenol, epidural bupivacaine
  * Postoperative: hydromorphone PCA, ibuprofen, oxycodone
  Interventions: Drug: Bupivacaine
- Intrathecal morphine with intraoperative lidocaine infusion (Experimental): * Day of surgery: tylenol, gabapentin, celebrex, and preoperative intrathecal morphine one time injection (150mcg)
  * Intraoperative: dexamethasone and lidocaine infusion 1 mg/kg ideal body weight
  * Day of surgery postoperative: toradol, ibuprofen, tylenol
  * Postoperative: ibuprofen, oxycodone, and hydromorphone prn
  Interventions: Drug: Morphine; Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine — -Epidural bupivacaine 0.1% 2-6ml/hr based on MAP within 10% of patient's baseline MAP
  Arms: Epidural bupivacaine with hydromorphone patient-controlled anesthesia (EPCA)
Drug: Morphine — -Preservative-free intrathecal morphine (duramorph) 150mcg injection (0.15ml or a 0.5mg/0.5ml prepared solution)
  Other Names: Duramorph
  Arms: Intrathecal morphine with intraoperative lidocaine infusion
Drug: Lidocaine — -Lidocaine infusion 1 mg/kg ideal body weight (IBW)
  Arms: Intrathecal morphine with intraoperative lidocaine infusion

SUMMARY:
To determine if opioid consumption postoperatively among patients undergoing non-emergent laparotomy by the gynecologic oncology service who receive intrathecal morphine with intraoperative lidocaine (IML) infusion are lower than patients who have epidural anesthesia with PCA (EPCA).

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years old
* Undergoing non-emergent exploratory laparotomy with the Gynecologic Oncology service
* No clinical or laboratory evidence of end organ failure:

If available:

* Platelets > 100 K/cumm
* Hemoglobin > 8.0 g/dl
* Serum creatinine <1.5 mg/dl
* Creatine clearance (CrCl) ≥30 based on the original Cockcroft-Gault formula adjusted for weight.
* INR <1.3 reference range
* All other lab values obtained as part of general preoperative work-up must be ≤1.5x normal laboratory value.

Exclusion Criteria:

* Patients not giving consent to participate in the study
* Unable to complete self-report pain questionnaire
* Moderate to severe kidney or liver failure per lab criteria as outlined
* Inability to hold anticoagulant medications for a safe amount of time per current ASRA guidelines
* Contraindication to lumbar puncture or epidural placement, per acute pain management service such as known coagulopathy or history of clotting disorders, history of scoliosis or lumbar fusion, infection at site of entry, or current systemic infection
* Complete bowel obstruction
* Contraindication to intravenous lidocaine
* No known pregnancy and not lactating.
* Currently septic
* Patient currently taking more than 30 MME a day preoperatively (for >30 days)
* BMI >50kg/m2
* Intolerance/contraindication or allergy to receiving non-steroidal anti-inflammatory drugs or acetaminophen or any other medications in the pre-operative order set

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premal H Thaker, M.D., MS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Started | 56 | 54
Completed | 50 | 46
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Determined to be ineligible | 0 | 1
Not completed — Withdrawn due to patient being given heparin | 0 | 1
Not completed — Technical failure | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Median (Full Range); unit: years] | 60 [23 to 82] | 64 [24 to 84] | 60 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 55 | 53 | 108
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 6 | 13
  White | 44 | 45 | 89
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 56 | 54 | 110

OUTCOME MEASURES:

1. Primary Outcome: Morphine Milligram Equivalent (MME) in the Postoperative Hospital Course
Time Frame: Postoperatively while patient is in hospital (estimated to be 4 days)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
mg | 89.9 (106.1) | 45.0 (89.8)
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.0249, Two-sample t-test; Unadjusted analysis; Mean Difference (Final Values) = -44.9, 95% CI 2-sided [-84.0 to -5.8] — Intrathecal - Epidural

2. Secondary Outcome: Rate of Postoperative Ileus
Description: Defined by bilious emesis requiring a change in diet to nothing-per-mouth (NPO) status or nasogastric tube placement (NGT) in the absence of other indications. Patients who had NGT placed prophylactically at the time of surgery were not considered to have an ileus unless an NGT was reinserted or they met the above criteria. Participants will be assigned a value of yes ileus or no ileus. The rate of post op ileus is defined as the observed number of yes ileus in each study arm divided by the total number of subjects in the study arm.
Time Frame: Postoperatively while patient is in hospital (estimated to be 4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
Participants | 6 | 6
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.94, Chi-squared; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.36 to 3.01] — Estimated probability of having the event in Intrathecal group divided by that in Epidural group

3. Secondary Outcome: Length of Hospital Stay
Description: Length of stay will be determined by the dates of admission as recorded in EPIC (days).
Time Frame: Estimated to be 4 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
days | 4.7 (2.0) | 4.4 (1.8)
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.59, Bootstrap resampling method; Bootstrap resampling method based on raw data was applied for due to highly right-skewed data (5,000 Bootstrap samples were selected); Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.01 to 0.48] — Intrathecal - Epidural

4. Secondary Outcome: Rate of Postoperative Hypotension
Description: -Postoperative hypotension will be defined as <90/50 (as previously defined by Huepenbecker, et al.) or a 20% decrease from the preoperative office visit.
Time Frame: Up to 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
Participants | 23 | 21
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.82, Chi-squared; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.61 to 1.48] — Estimated probability of having the event in Intrathecal group divided by that in Epidural group

5. Secondary Outcome: Patient Satisfaction With Pain Control
Description: -Patients will be asked on day of discharge if they were satisfied with their pain control during their hospitalization. They will be able to choose from the following: 0=satisfied, 1= somewhat satisfied, 2= neutral, 3=somewhat dissatisfied, 4=dissatisfied).
Time Frame: Day of hospital discharge (estimated to be day 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
Participants
  Very satisfied | 41 | 42
  A little satisfied | 8 | 5
  Not sure | 0 | 2
  A little dissatisfied | 1 | 0
  Very dissatisfied | 1 | 0

6. Secondary Outcome: Change in Pain Scores
Description: Pain scores will be determined by the 0-10 numeric rating scale (NRS). 0=no pain and 10=the most pain. A higher score indicates more pain.
Time Frame: Preoperative, each post-operative day while inpatient, 2 week follow-up, and 6 week follow-up
Population: The number analyzed at the different time points may be different than the overall number analyzed due to participant not being hospitalized at the time point or the pain score not being completed at the time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
score on a scale
  Preoperative | 1.7 (2.3) | 1.7 (2.2)
  Day of surgery | 3.7 (2.1) | 2.0 (1.8)
  Post-operative day 1 | 3.7 (2.3) | 3.0 (2.1)
  Post-operative day 2 | 3.7 (2.4) | 3.3 (2.1)
  Post-operative day 3: number analyzed (Participants) | 33 | 32
  Post-operative day 3 | 3.3 (2.3) | 2.8 (1.9)
  Post-operative day 4: number analyzed (Participants) | 17 | 11
  Post-operative day 4 | 3.3 (2.3) | 2.9 (1.9)
  Post-operative day 5: number analyzed (Participants) | 13 | 9
  Post-operative day 5 | 3.0 (2.7) | 2.6 (2.3)
  Post-operative day 6: number analyzed (Participants) | 10 | 8
  Post-operative day 6 | 2.5 (1.9) | 2.3 (2.8)
  Post-operative day 7: number analyzed (Participants) | 6 | 4
  Post-operative day 7 | 1.9 (2.1) | 2.0 (3.6)
  Post-operative day 8: number analyzed (Participants) | 4 | 2
  Post-operative day 8 | 2.1 (2.5) | 3.3 (4.6)
  Post-operative day 9: number analyzed (Participants) | 1 | 2
  Post-operative day 9 | 4.8 | 3.3 (3.9)
  Post-operative day 10: number analyzed (Participants) | 0 | 0
  2 week follow-up: number analyzed (Participants) | 50 | 48
  2 week follow-up | 1.9 (1.8) | 1.6 (1.7)
  6 week follow-up: number analyzed (Participants) | 46 | 45
  6 week follow-up | 0.85 (1.5) | 0.76 (1.7)

7. Secondary Outcome: 30 Day Readmission Rate
Time Frame: Through day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
Participants | 2 | 3
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.67, Fisher Exact; Risk Ratio (RR) = 1.56, 95% CI 2-sided [0.27 to 8.95] — Estimated probability of having the event in Intrathecal group divided by that in Epidural group

8. Secondary Outcome: Rate of Deep Vein Thrombosis (DVT) or Pulmonary Thromboembolism (PTE)
Time Frame: From day of surgery (day 1) to 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 51 | 49
Participants | 1 | 2
Statistical Analysis 1: Comparison: Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) vs Intrathecal Morphine With Intraoperative Lidocaine Infusion; Test type: Superiority; p = 0.61, Fisher Exact; Risk Ratio (RR) = 2.08, 95% CI 2-sided [0.19 to 22.2] — Estimated probability of having the event in Intrathecal group divided by that in Epidural group

9. Secondary Outcome: Rate of Persistent Pain
Description: -As determined by an NRS pain score ≥ 5
Time Frame: At 6 week follow-up
Population: Only participants who had the NRS Pain Score at 6 week follow-up are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
Number analyzed (Participants) | 46 | 45
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from day of surgery through 6-week follow-up.
Arm/Group | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) | Intrathecal Morphine With Intraoperative Lidocaine Infusion
All-Cause Mortality (participants affected / at risk) | 0/51 | 2/49
Serious Adverse Events (participants affected / at risk) | 6/51 | 4/49
Other Adverse Events (participants affected / at risk) | 36/51 | 41/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) (N=51) | Intrathecal Morphine With Intraoperative Lidocaine Infusion (N=49)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 | 0
Hypovolemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Death due to endometrial cancer (General disorders) | 0 | 1
Generalized edema (General disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Adult respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Surgery (exploratory laparotomy/large bowel resection/end colostomy/mucous fistula procedure) (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural Bupivacaine With Hydromorphone Patient-controlled Anesthesia (EPCA) (N=51) | Intrathecal Morphine With Intraoperative Lidocaine Infusion (N=49)
Anemia (Blood and lymphatic system disorders) | 6 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 1 | 1
Fever (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Intestinal stoma obstruction (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Creatinine increased (Investigations) | 10 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 8
Prerenal acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urine output decreased (Renal and urinary disorders) | 1 | 2
Genital edema (Reproductive system and breast disorders) | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Delayed awakening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 22 | 19
Thromboembolic event (Vascular disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT05017246/Prot_SAP_000.pdf